CLINICAL TRIAL: NCT01226810
Title: A Novel Approach to Ultrafast Parathyroid SPECT Imaging Using a Solid State CZT SPECT Camera
Brief Title: The Novel Approach of Minimally Invasive Parathyroid Surgery Requires Precise Identification and Localization of the Lesion Prior to Exploration
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Prof. Ora Israel, RambamMC
Other Study IDs: 024-10-RMB_parathyroid
Record Dates: First submitted 2010-10-21; First posted 2010-10-22 (Estimated); Last update posted 2010-10-22 (Estimated); Status verified 2010-10

CONDITIONS: Hypercalcemia; Hyperparathyroidism
MeSH Terms: conditions — Hypercalcemia; Hyperparathyroidism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Purpose of this study is to compare the image quality and diagnostic accuracy obtained with ultrafast solid state short SPECT in comparison with the routine SPECT protocol.

DETAILED DESCRIPTION:
Single-tracer, dual-phase Tc-MIBI parathyroid scintigraphy is based on the differential washout rate of the tracer (MIBI) from the thyroid and the parathyroid tissue. A distinct focus of increased MIBI uptake relative to the thyroid gland, either on the early or late image or on both, or a focal uptake in the mediastinum, is considered positive for abnormal parathyroid tissue. Tc99m-MIBI planar scintigraphy was found to play a major role in the preoperative localization of a parathyroid adenoma (PTA), with a sensitivity ranging from 85% to 95% and specificity of up to 99%. Subsequently, the use of MIBI- Single photon emission computed tomography (SPECT) significantly improved the sensitivity of the test and improved the accuracy of lesion localization.

A limitation of adding the SPECT component is related to its relatively long duration. The duration of a MIBI-SPECT acquisition of neck and the mediastinal area may take up to 15-20 minutes using a standard nuclear medicine camera. Long acquisition time may lead to patient discomfort and movement resulting in image degradation, artifacts and may lead to overall decreased diagnostic accuracy.

A reduced SPECT acquisition time without image quality degradation may decrease patient discomfort and increase clinical throughput. An ultrafast solid state CZT camera (GE Healthcare Discovery 570C) is currently used for routine cardiac SPECT imaging achieving high quality cardiac studies for a significantly shorter acquisition time. Present study evaluates the potential use of the ultrafast camera in patients with a clinically suspected PTA who perform Tc-MIBI imaging.

ELIGIBILITY:
Inclusion Criteria:

1) The subject is 18 years old or older. (2) The subject is clinically suspected or known to have parathyroid adenoma and is scheduled to have a MIBI study as part of his/her standard clinical evaluation.

(3) The subject is able and willing to comply with the additional procedure (ultrafast MIBI SPECT) and a signed and dated informed consent is obtained before any procedure for study purposes is performed.

Exclusion Criteria:

1. Pregnancy.
2. Psychosis or any other condition, which, in the investigators opinion would prevent adherence to the study protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for the parathyroid scan.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-01

CONTACTS AND LOCATIONS:
Overall Officials: Ora Israel, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Healthcare Campus, Haifa, Israel

REFERENCES:
- [Derived] Chen J, Gopala K, Akarsh PK, Struyf F, Rosillon D. Prevalence and Incidence of Human Papillomavirus (HPV) Infection Before and After Pregnancy: Pooled Analysis of the Control Arms of Efficacy Trials of HPV-16/18 AS04-Adjuvanted Vaccine. Open Forum Infect Dis. 2019 Dec 4;6(12):ofz486. doi: 10.1093/ofid/ofz486. eCollection 2019 Dec. PMID 31824976
- [Derived] Safaeian M, Castellsague X, Hildesheim A, Wacholder S, Schiffman MH, Bozonnat MC, Baril L, Rosillon D; Costa Rica HPV Vaccine Trial and the PATRICIA study groups. Risk of HPV-16/18 Infections and Associated Cervical Abnormalities in Women Seropositive for Naturally Acquired Antibodies: Pooled Analysis Based on Control Arms of Two Large Clinical Trials. J Infect Dis. 2018 Jun 5;218(1):84-94. doi: 10.1093/infdis/jiy112. PMID 29718393